CLINICAL TRIAL: NCT00001872
Title: Apheresis of Family Members of Patients Undergoing Allogeneic Bone Marrow Transplantation. A Pre-Clinical Study of Selective Depletion of Donor Lymphocytes to Prevent Acute Graft-Versus-Host Disease
Brief Title: Cell Selection for Bone Marrow Transplants to Prevent Graft-Versus-Host-Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990037; 99-H-0037
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-03-02

CONDITIONS: Graft vs Host Disease; Hematologic Neoplasm
Keywords: Volunteer; Leukocyte Donors; Family Members; Leukocyte Collection; No Reimbursement
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Blood contains different kinds of cells, white blood cells, red blood cells, and platelets. In order to treat certain diseases, specific cell types can be removed from blood and transplanted into patients. The process of removing white blood cells for the treatment of leukemia is called apheresis.

This study will make available blood cell collections from volunteers genetically matched to various degrees with recipients in order to test and, if necessary, refine the process of removing white blood cell T-lymphocytes....

DETAILED DESCRIPTION:
This protocol has been written to make available apheresis collections from volunteers matched to various degrees with recipients in order to test and, if necessary refine, the selective immunodepletion procedure prior to introducing it in a clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Family members of patients admitted to NHLBI allogeneic BMT protocols.

Ages 18 and older and less than age 65.

Parent of patient (obligate haplotype match) OR HLA 3/6, 4/6, 5/6, or 6/6 match with patient.

Research apheresis available from patient.

EXCLUSION CRITERIA:

Pregnancy or lactation.

HLA type unknown.

More than one haplotype mismatch with patient.

History of any immunosuppressive disease.

History of chronic viral antigenic stimulus.

Venous access inadequate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1999-02-02; Study Completion 2018-03-02

CONTACTS AND LOCATIONS:
Overall Officials: A. John Barrett, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Datta AR, Barrett AJ, Jiang YZ, Guimaraes A, Mavroudis DA, van Rhee F, Gordon AA, Madrigal A. Distinct T cell populations distinguish chronic myeloid leukaemia cells from lymphocytes in the same individual: a model for separating GVHD from GVL reactions. Bone Marrow Transplant. 1994 Oct;14(4):517-24. PMID 7858526
- [Background] Mavroudis DA, Jiang YZ, Hensel N, Lewalle P, Couriel D, Kreitman RJ, Pastan I, Barrett AJ. Specific depletion of alloreactivity against haplotype mismatched related individuals by a recombinant immunotoxin: a new approach to graft-versus-host disease prophylaxis in haploidentical bone marrow transplantation. Bone Marrow Transplant. 1996 May;17(5):793-9. PMID 8733700
- [Background] Mavroudis DA, Dermime S, Molldrem J, Jiang YZ, Raptis A, van Rhee F, Hensel N, Fellowes V, Eliopoulos G, Barrett AJ. Specific depletion of alloreactive T cells in HLA-identical siblings: a method for separating graft-versus-host and graft-versus-leukaemia reactions. Br J Haematol. 1998 Jun;101(3):565-70. doi: 10.1046/j.1365-2141.1998.00748.x. PMID 9633903